CLINICAL TRIAL: NCT07168525
Title: Effects of Ultrasound on Healthy Aging
Brief Title: Ultrasound for Healthy Aging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Xprize Foundation (Unknown)
Responsible Party: Principal Investigator, Blake Rasmussen, Professor and Chairman of Dept. of Cellular & Integrative Physiology, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00001878
Record Dates: First submitted 2025-08-26; First posted 2025-09-11 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-08

CONDITIONS: Aging
Keywords: Ultrasound; Muscle function; Cognitive function
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Randomized controlled 2 arm study
Who Masked: Participant
Masking Description: This sham-controlled design improves internal validity by minimizing placebo effects and allows for participant blinding, as the ultrasound is inaudible and imperceptible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Ultrasound Spa Group (Experimental): Sessions will take place three times per week, with water-based delivery of low-frequency ultrasound lasting 45 minutes each, for a total of eight weeks.
  Interventions: Device: Ultrasound spa
- Spa Only Group without ultrasound (Sham Comparator): Sessions will take place three times per week, with spa immersion with no ultrasound lasting 45 minutes each, for a total of eight weeks.
  Interventions: Other: Sham ultrasound spa

INTERVENTIONS:
Device: Ultrasound spa — Each participant will sit in a bathtub which has been fitted with an ultrasound device which produces low frequency sound waves within the water.
  Other Names: Bathtub with ultrasound
  Arms: Ultrasound Spa Group
Other: Sham ultrasound spa — The control group will sit in the same tub for 45 minutes, 3 times per week for 8 weeks but without the ultrasound being turned on.
  Other Names: Bathtub with ultrasound deactivated
  Arms: Spa Only Group without ultrasound

SUMMARY:
The investigators will study the effects of an ultrasound bath device that uses low-frequency ultrasound on the healthy aging. Participants will have before and after ultrasound assessments of muscle and thinking skills, aging related to the immune system, and body make-up. The group that is assigned to get the ultrasound will have low-frequency ultrasound in a bathtub for 45 minutes, three times weekly for 8 weeks, and the control group will be in the bathtub without the ultrasound turned on.

DETAILED DESCRIPTION:
The general approach and study design is that the investigators will recruit 20 healthy older adults (equal numbers of men and women) for the first phase. 10 participants will be randomized to the ultrasound group and 10 will be randomized to the control group. Participants will be stratified by gender and ten randomized to treatment arms. Prior to beginning the intervention, each participant will be tested for muscle function, cognitive function, blood samples will be used to assess immune aging function, and body composition. Each participant will then sit in a bathtub which has been fitted with an ultrasound device which produces low frequency sound waves within the water. The sound waves are undetectable by someone sitting in the tub. The ultrasound intervention group will receive ultrasound for 45 minutes, 3 times per week for 8 weeks. The control group will sit in the same tub for 45 minutes, 3 times per week for 8 weeks but without the ultrasound being turned on. At the end of the 8 weeks, post-testing for muscle, cognitive, immune aging function, and body composition will be performed again.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females; Age 70 or older
2. BMI <40 kg/m2
3. Ability to walk up a flight of stairs and short ladder
4. Ability to get in and out of a bath
5. Willingness to adhere to the spa treatments regimen

Exclusion Criteria:

1. To accommodate the participants comfortably in our spa, participants with body weight >350 pounds, body girth ≥ 50 inches and height ≥ 6 feet 8 inches will be excluded.
2. Any medical condition that, in the opinion of the investigator, would place the participant at increased risk for participation.
3. Fecal or urinary incontinence (daily use of depends)
4. Uncontrolled HTN (BP >180) or unstable vital signs that in the opinion of the investigator would place at increased risk for participation
5. Any clinically significant rash or formation of rashes or open sores, boils, or infected wounds two weeks prior to screening or any time during the study.
6. History of poor wounds healing lower extremity within the past two years
7. Glycated Hemoglobin (Hgb) A1c level >8.5%
8. Required use of ambulatory assistive devices
9. Laboratory evidence of infection or colonization with multidrug resistant pathogens in the past 90 days
10. History of myocardial infarction (MI), cerebrovascular accident (CVA) within the past year
11. History of prior non-compliance or the presence of history of health condition (drug or alcohol addiction) that would make it difficult for the participant to comply with the study procedures or follow the investor's instructions
12. Unable to complete procedures in visit 1

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee Extension Strength change | Baseline to 8 weeks
  A sensitive and reliable measure of lower-extremity muscle function andis clinically relevant for predicting mobility limitations and fall risk in older adults measured by Biodex dynamometry.

SECONDARY OUTCOMES:
Change in Short Physical Performance Battery (SBBP) | Baseline to 8 weeks
  A well-established objective measure of lower extremity physical function that includes balance testing, timed 4 meter walk, and timed repeated chair stands.Scores for each test are graded on a 0-4 scale and the total for each test summed to provide a total between 0-12 where 0 is the worst performance and 12 is the best.
Change in Timed Up and Go (TUG) | Baseline to 8 weeks
  The Timed Up and Go (TUG) test is a simple assessment used to evaluate a person's functional mobility and risk of falls, particularly in older adults. The test involves timing how long it takes for an individual to stand up from a chair, walk a short distance, turn around, walk back, and sit down again.
Change in 6 minute walk distance | Baseline to 8 weeks
  Will measure the maximal distance participants can walk during six minutes. Participants will be instructed to "cover as much distance as they can" over a flat surface demarcated by traffic cones while timed by a stopwatch.
Change in Senescence | Baseline to 8 weeks
  Cellular senescence in blood will be measured via immunohistochemistry biochemical analysis and RNA sequencing.
Change in immune aging | Baseline to 8 weeks
  Immune aging in blood will be measured via epigenetic analysis.
Change in cognitive function | Baseline to 8 weeks
  Cognitive function will be measured via the NIH Toolbox Cognition Battery Face Name Associative Memory Exam Test. Participants will be shown 12 pairs of names and faces followed by a 5-25 minute break prior to being shown the pairs again. The possible scores are 0-12. 0 is no names and faces remembered and 12 is all pairs remembered correctly.
Change in lean body mass | Baseline to 8 weeks
  Measured by a DEXA scan
Change in fat mass | Baseline to 8 weeks
  Measured by DEXA scan

CONTACTS AND LOCATIONS:
Overall Officials: Blake Rasmussen, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will ensure all mechanisms used to share data will include proper plans and safeguards for the protection of privacy, confidentiality, and security for data dissemination and reuse (e.g., all data will be thoroughly de-identified and will not be traceable to a specific study participant). Plans for archiving and long-term preservation of the data will be implemented, as appropriate.
Supporting Information: Study Protocol, SAP
Time Frame: At study completion at the time of publication in a peer review journal